CLINICAL TRIAL: NCT04509141
Title: Acupuncture as Migraine Prophylaxis in Reducing Frequency, Duration and Intensity of Migraine With Minimum Acupoint, Seen up to Eight Weeks From Baseline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Newanda Johni Muchtar, Sp. Ak, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: medical acupuncture 2020
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Migraine; Headache; Migraine Disorders
Keywords: migraine; acupuncture; visual analogue scale; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with control was conducted on 34 subjects with migraine who were randomly allocated into the manual group of acupuncture (n = 17), as well as the medicine group (n = 17). The assessment of frequency, duration and intensity of migraine attacks assessed at the time before treatment, at the fourth and eight week from baseline
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the patient did not know that there were two groups divided in each participants, and the doctor who measures the outcome also did not know which person belongs to which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupuncture (Active Comparator): acupuncture three times a week
  Interventions: Other: acupuncture
- standard treatment for migraine by neurologist (Active Comparator): standard treatment for migraine that was given by a neurologist
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — acupuncture points used were EXHN5 Taiyang, GB20 Fengchi, TE5 Waigun, GB41 Zulinqi

SUMMARY:
Migraine is a primary headache attack, specific, paroxysmal, with or without aura, with subjective manifestations both before and after the attack, a chronic type of headache with symptoms of recurrence, attacks at productive age and can cause a decrease in work productivity up to 80%, so that it will affect the quality of life, economic life and education globally which leads to losses for migraine sufferers and institutions where migraine sufferers attend school, work and in the lives of sufferers' families.

DETAILED DESCRIPTION:
Migraine is a primary headache attack, specific, paroxysmal, with or without aura, with subjective manifestations both before and after the attack, a chronic type of headache with symptoms of recurrence, attacks at productive age and can cause a decrease in work productivity up to 80%, so that it will affect the quality of life, economic life and education globally which leads to losses for migraine sufferers and institutions where migraine sufferers attend school, work and in the lives of sufferers' families. With the high prevalence and disability rates for migraine sufferers, on the other hand, the right treatment for migraine has not yet been obtained to the maximum, it is necessary to deepen the treatment and prevention of migraine is needed, and until now there has been no definitive cure, both for prevention and treatment, so it is necessary to develop therapies that can provide more accurate relief for migraine sufferers. The purpose of this study is to assess the success in managing migraine in reducing the frequency of attacks, reducing the intensity of attacks and reducing the duration of attacks from weeks 0, 4 to 8

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 19-50 years
* subjects with history of clinical diagnosis of migraine (interictal period)
* signed research approval forms, and were willing to take the study to completion.

Exclusion Criteria:

* subjects with pregnancy,
* lesions, wounds, infections and suffering from malignant diseases or tumor and thrombophlebitis in the area at the selected acupuncture point
* increasing liver function three times above normal values.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
frequency | at week 4
  Manual acupuncture interventions can reduce the frequency of migraine attacks better than the preventive pharmacological valproic acid
duration | at week 4
  Manual acupuncture interventions can reduce the duration of migraine attacks better than the preventive pharmacological valproic acid
intensity | at week 4
  Manual acupuncture interventions can reduce the change from Baseline in pain scores on the Visual Analog Scale of migraine attacks better than the preventive pharmacological valproic acid
frequency | at week 8
  Manual acupuncture interventions can reduce the frequency of migraine attacks better than the preventive pharmacological valproic acid
duration | at week 8
  Manual acupuncture interventions can reduce the duration of migraine attacks better than the preventive pharmacological valproic acid
intensity | at week 8
  Manual acupuncture interventions can reduce the change from Baseline in pain scores on the Visual Analog Scale of migraine attacks better than the preventive pharmacological valproic acid

CONTACTS AND LOCATIONS:
Locations (1):
- University of Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia